CLINICAL TRIAL: NCT04933864
Title: The Clinical Trial of Methylene Blue Application Combined With Photodynamic Therapy for Treatment of SARS-CoV-2 Infected Patients
Brief Title: COVID-19 Treatment Using Methylene Blue and Photodynamic Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Collaborators: Prokhorov General Physics Institute of the Russian Academy of Sciences (GPI RAS) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2206
Record Dates: First submitted 2021-06-15; First posted 2021-06-22 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: SARS-CoV-2
Keywords: COVID-19; photodynamic therapy; methylene blue
MeSH Terms: conditions — COVID-19 | interventions — Methylene Blue; Photochemotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methylene Blue and Photodynamic Therapy (Experimental): Methylene Blue 1 mg/kg water solution. Participants have orally received Methylene Blue solution of 1 mg/kg concentration one time in addition to the current therapy of the participant (e.g., azithromycin, hydroxychloroquine, aminodihydrophthalazinedione sodium, levofloxacin, etc.), if any. After 3 hours of Methylene Blue administration irradiation of chest using 650 nm laser source with 18 J/cm^2 energy dose was performed.
  Interventions: Drug: Methylene Blue and Photodynamic Therapy
- Control group (No Intervention): COVID-19 positive participants treated with standard medical supportive therapy (e.g. azithromycin, hydroxychloroquine, aminodihydrophthalazinedione sodium, levofloxacin, etc.).

INTERVENTIONS:
Drug: Methylene Blue and Photodynamic Therapy — Treatment group. Methylene blue (SamaraMedProm, Russia, Registration number: MP-001834, 13.09.2012) 1 mg/kg concentration orally one time were added to the current therapy of the participant (e.g., azithromycin, hydroxychloroquine, aminodihydrophthalazinedione sodium, levofloxacin, etc.), if any, and irradiation of the participant's chest was performed by 650 nm laser source (UFPh-675-01-BIOSPEC, BIOSPEC, Russia, Registration number: 2009/04648, 26.03.2009) with 18 J/cm^2 energy dose.
  For critically ill participants: Inhalation by 0.2 mg methylene blue (SamaraMedProm, Russia, Registration number: MP-001834, 13.09.2012) 10 ml water solution and irradiation of pharynx and nasal cavity by 650 nm laser source (UFPh-675-01-BIOSPEC, BIOSPEC, Russia, Registration number: 2009/04648, 26.03.2009) with 36 J/cm^2 energy dose were performed.
  Other Names: Methylene Blue (SamaraMedProm, Russia, Registration number: MP-001834, 13.09.2012), 650 nm laser source (UFPh-675-01-BIOSPEC, BIOSPEC, Russia, Registration number: 2009/04648, 26.03.2009)
  Arms: Methylene Blue and Photodynamic Therapy

SUMMARY:
According to the epidemiological situation worldwide and the number of vaccinations made, there is little success in the fight against COVID-19. For many reasons, methylene blue is a promising drug for an active treatment against SARS-CoV-2 infected patients. Since methylene blue can work as a photosensitizer, photodynamic therapy as an antiviral treatment has great potential in the treatment of COVID-19. This clinical study investigated the effectiveness of SARS-CoV-2 infected people treatment using methylene blue and the following photodynamic therapy on the base of the L.L. Levshin Institute of Cluster Oncology (Department of Infectious Diseases №13) of I.M. Sechenov First Moscow State Medical University.

DETAILED DESCRIPTION:
This is a randomized, parallel, single masking clinical study 60 participants aged 18-90 with one positive COVID-19 quantitative Polymerase Chain Reaction test and any severity of pneumonia (checked by computer tomography scans) were recruited. The experimental and control samples included 30 participants. Randomization was performed using the Random Number Table generated in STATISTICA Advanced 13.3. The physiological parameters including oxygen saturation, severity of pneumonia using computer tomography scans, heart rate, symptoms, and physical examination were collected. Participants in the experimental sample received methylthioninium chloride, Methylene Blue (SamaraMedProm, Russia, Registration number: MP-001834, 13.09.2012) orally in concentration 1 mg/kg in addition to the current therapy of the participant (e.g., azithromycin, hydroxychloroquine, aminodihydrophthalazinedione sodium, levofloxacin, etc.), if any. After 3 hours, photodynamic therapy of the participant's chest by a 650 nm laser source (UFPh-675-01-BIOSPEC, BIOSPEC, Russia, Registration number: 2009/04648, 26.03.2009) with 18 J/cm^2 energy dose was performed for 50 minutes. If the participant is in a critical state, inhalation by 0.2 mg Methylene Blue 10 ml water solution and following photodynamic therapy of pharynx and nasal cavity using 650 nm laser source with 36 J/cm^2 energy dose during 10 minutes were performed. Participants in the control sample received only standard medical supportive therapy (e.g., azithromycin, hydroxychloroquine, aminodihydrophthalazinedione sodium, levofloxacin, etc.). All next steps were performed for p participants from the experimental sample: 12 and 24 hours after photodynamic therapy, blood saturation were measured. 2 days after - participants will take a quantitative polymerase chain reaction test. 14 days after - computer tomography Aquilion One 640 (Canon Medical Systems Corporation, Registration Certificate FSZ 2008/01304, 02.07.2018) scans were performed. The participant's status scale (EQ-5D-3L, SHOCS-COVID score, validated) was checked on day 84. On 24 and 84 days all participants were checked whether they are alive or not by phone call. For participants in the control sample continuous check of blood saturation, quantitative Polymerase Chain Reaction tests after 2 and 14 days of treatment, and computer tomography scans were performed. The primary outcome of this study is to calculate the percentage of participants with negative quantitative Polymerase Chain Reaction test on SARS-CoV-2 by 2 days after methylene blue administration and photodynamic therapy. Experimental and control samples were comparable in gender, age, and severity of the disease. Z-test was used to analyze results on quantitative Polymerase Chain Reaction tests within control and experimental samples. For each sample paired Student t-test was used to analyze individual saturation changes. Wilcoxon criterion was used for data on severity of pneumonia and status scale.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* age: 18-90 years
* positive quantitative Polymerase Chain Reaction test on SARS-CoV-2 infection
* negative pregnancy test in women
* any severity of pneumonia (computer tomography scans)

Non-inclusion Criteria:

* documented refusal to participate in the study
* treatment with a serotonergic drug
* connection to artificial lung ventilation with or without sedation
* history of G-6-Phosphatase deficiency
* pregnancy and breastfeeding
* medical records of cirrhosis
* active chronic hepatitis

Exclusion Criteria:

* myocardial infarction, developed after the patient was included in the study, but before the intervention
* bleeding, developed after the patient was included in the study, but before the intervention
* connection to artificial lung ventilation developed after the patient was included in the study, but before the intervention

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-04-24 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
The percentage of participants with negative quantitative Polymerase Chain Reaction test on SARS-CoV-2 on day 2 after methylene blue administration and photodynamic therapy | Day 2
  The percentage of participants with negative quantitative Polymerase Chain Reaction test was reported. Quantitative Polymerase Chain Reaction test was performed not earlier than 3-4 hours after the last meal, excluding the use of medicines for topical application (drops, sprays, etc.) before taking the test.

SECONDARY OUTCOMES:
Comparison of oxygen saturation dynamics measured by pulse oximeter before and after treatment | 12 and 24 hours after photodynamic therapy
  The saturation dynamics after photodynamic therapy in 12 and 24 hours were reported
The percentage of participants with positive dynamics in severity of pneumonia (e.g., from CT-4 to CT-2) | Day 14
  The percentage of participants that have a positive trend in severity of pneumonia (computer tomography scans) after treatment (e.g., from CT-4 to CT-2) was reported
The percentage of participants having positive dynamics in patient status scale (EQ-5D-3L, SHOCS-COVID score) after treatment | Day 84
  The percentage of participants that have positive dynamics in patient status scale (EQ-5D-3L, SHOCS-COVID score) was calculated
The percentage of participants alive at day 28 | Day 28
  The percentage of participants still alive at day 28 of samples collection was reported
The percentage of participants alive at day 84 | Day 84
  The percentage of participants still alive at day 84 of samples collection was reported

CONTACTS AND LOCATIONS:
Overall Officials: Igor V. Reshetov, Prof., Study Director — I.M. Sechenov First Moscow State Medical University (Sechenov University); Artem A. Shiryaev, Ph.D., Principal Investigator — I.M. Sechenov First Moscow State Medical University (Sechenov University); Victor B. Loschenov, Prof., Study Chair — Prokhorov General Physics Institute of the Russian Academy of Sciences
Locations (1):
- I.M. Sechenov First Moscow State Medical University (Sechenov University), Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
The Local Ethics Committee of I.M. Sechenov First Moscow State Medical University did not give permission to provide individual participant data.

REFERENCES:
- [Background] Strakhovskaya, M. G., Meerovich, G. A., Kuskov, A. N., Gonchukov, S. A., & Loschenov, V. B. (2020, September 1). Photoinactivation of coronaviruses: Going along the optical spectrum. Laser Physics Letters. IOP Publishing Ltd. https://doi.org/10.1088/1612-202X/abab14